CLINICAL TRIAL: NCT00442325
Title: ACTFAST (2): Achieve Cholesterol Targets Fast With Atorvastatin Stratified Titration: A Multicenter, Twelve-Week Treatment, Single-Step Titration, Open-Label Study Assessing The Percentage Of Dyslipidemic High-Risk Patients Achieving Low Density Lipoprotein Cholesterol (LDL-C) Target With Atorvastatin Starting Doses Of 10 mg, 20 mg, 40 mg, And 80 mg.
Brief Title: Benefits Of Using Various Starting Doses Of Atorvastatin On Achievement Of Cholesterol Targets
Acronym: ACTFAST 2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2581095
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Coronary Arteriosclerosis; Diabetes Mellitus, Type 2; Cerebrovascular Accident; Dyslipidemia; Peripheral Vascular Disease
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus, Type 2; Stroke; Dyslipidemias; Peripheral Vascular Diseases | interventions — Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin (Lipitor)

SUMMARY:
European physicians tend to always use the lowest dose of statins to initiate therapy even in subjects who require large reductions in cholesterol. The study evaluates if selecting the starting dose based on baseline and target LDL-C cholesterol would provide better results (ie proportion of subjects resching target)

ELIGIBILITY:
Inclusion Criteria:

* High cholesterol blood levels (LDL-cholesterol above 100 mg/dL up to 220 mg/dL.
* Triglycerides up to 600 mg/dL.
* History of coronary artery disease (ex.: heart attack, angina), stroke, diabetes or at high risk of such events.

Exclusion Criteria:

* Pregnancy or lactation, use of high statin doses (>40mg) at baseline, liver or renal problems
* Use of other drugs that would interfere with evaluation of efficacy or cause safety problems
* Uncontrolled hypertension, diabetes or hypothyroidism
* Recent cardiac event of procedure
* High baseline CPK levels

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 595
Dates: Start 2003-01; Study Completion 2004-02

PRIMARY OUTCOMES:
Proportion of subjects achieving a LDL-C target of < 100 mg/dL (2.6 mmol/L) after 12 weeks.

SECONDARY OUTCOMES:
Percentage of subjects achieving:
LDL-C target <100 mg/dL (<2.6 mmol/L) after 6 weeks of treatment.
Total cholesterol (TC)/HDL-C ratio target (<4.0) after 6 and 12 weeks of treatment.
Either the LDL-C <100mg/dL (<2.6 mmol/L) or TC/HDL-C ratio (<4.0) targets after 6 and 12 weeks of treatment.
Both the LDL-C <100mg/dL (<2.6 mmol/L) and TC/HDL-C ratio (<4.0) targets after 6 and 12 weeks of treatment.
LDL-C <100mg/dL (<2.6 mmol/L) or TC/HDL-C ratio (<4.0) targets after 6 and 12 weeks of treatment by LDL-C strata.
LDL-C target (<100 mg/dL) by primary inclusion diagnosis (CHD, CHD-equivalent, diabetes or 10-year CHD risk-equivalent >20%).
The mean percent change in LDL-C, high density lipoprotein cholesterol (HDL-C),TC/HDL-C ratio, non HDL-C (in subjects with triglycerides [TG] ≥200 mg/dL or 2.3 mmol/L), TC and TG from baseline to 6 and 12 weeks of treatment. Change from baseline in apol

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (32):
- Greece (4):
  - Pfizer Investigational Site, Ioannina
  - Pfizer Investigational Site, Kallithea, Athens
  - Pfizer Investigational Site, Pireaus
  - Pfizer Investigational Site, Thessaloniki
- Hungary (5):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Gyula
  - Pfizer Investigational Site, Kecskemét
  - Pfizer Investigational Site, Nyíregyháza
  - Pfizer Investigational Site, Szekszárd
- Ireland (6):
  - Pfizer Investigational Site, Tullamore, CO. Offlay
  - Pfizer Investigational Site, Tallaght, Dublin
  - Pfizer Investigational Site, Gorey, Wexford
  - Pfizer Investigational Site, Cork
  - Pfizer Investigational Site, Dublin
  - Pfizer Investigational Site, Galway
- Poland (5):
  - Pfizer Investigational Site, Częstochowa
  - Pfizer Investigational Site, Poznan
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Wroclaw
  - Pfizer Investigational Site, Zabrze
- Portugal (4):
  - Pfizer Investigational Site, Aveiro
  - Pfizer Investigational Site, Lisbon
  - Pfizer Investigational Site, Porto
  - Pfizer Investigational Site, Vila Franca de Xira
- Pfizer Investigational Site, Moscow, Russia
- Slovakia (2):
  - Pfizer Investigational Site, Bratislava
  - Pfizer Investigational Site, Košice
- Switzerland (4):
  - Pfizer Investigational Site, Bern
  - Pfizer Investigational Site, Geneva
  - Pfizer Investigational Site, Mendrisio
  - Pfizer Investigational Site, Zurich
- Pfizer Investigational Site

REFERENCES:
- [Derived] Farsang C, Athyros V, Gaw A; ACTFAST-2 investigators and Steering Committee members. A multicentre, open study to assess the effect of individualizing starting doses of atorvastatin according to baseline LDL-C levels on achieving cholesterol targets: the Achieve Cholesterol Targets Fast with Atorvastatin Stratified Titration (ACTFAST-2) study. Curr Med Res Opin. 2007 Aug;23(8):1945-56. doi: 10.1185/030079907X223242. PMID 17626713
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581095&StudyName=Benefits+Of+Using+Various+Starting+Doses+Of+Atorvastatin+On+Achievement+Of+Cholesterol+Targets+%28ACTFAST+2%29